CLINICAL TRIAL: NCT01152567
Title: Effects of Angiotensin Converting Enzyme Inhibitors vs Candesartan in Reducing Cardiovascular Events in Primary Treatment of Hypertension
Brief Title: Effects of Angiotensin Converting Enzyme (ACE) Inhibitors Versus Candesartan in Reducing Cardiovascular Events in Primary Treatment of Hypertension
Acronym: ARBACE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CSE-ATA-2010/1
Record Dates: First submitted 2010-06-18; First posted 2010-06-29 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension; Cardiovascular Disease
Keywords: Hypertension; ACE; ARB; real life data; CVD; cost effectiveness
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACE: Patients treated for hypertension with ACEs without CVD
- Candesartan: Patients treated for hypertension with candesartan without CVD

SUMMARY:
The planned Study will be a retrospective study on the effect of ACE's vs. candesartan on cardiovascular events and on health economic effects in a "real life" setting in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* all patients found in electronic patient journals at the participating centres, who were prescribed either ACEis (ATC-C09A-B) or ARBs (C09C-D) for hypertension from 1 January 1999 - 31 December 2007. The first date of such a prescription starts the observation time and is called the index prescription.

Exclusion Criteria:

* No history of cardiovascular disease.
* Ongoing malignancy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient treated with ACE or candesartan in the period 1999 - 2007.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Investigate the risk of Cardiovascular Disease (CVD) and new onset diabetes in patients on primary hypertensive treatment with ACE or candesartan for hypertension | Time to first CV event calculated as the time (in days) between date of index prescription and date of the first registration of a CV event. Patients will be followed for min. 1 wk and up to 9 yrs (1999-2007). Median follow up time is estimated to 2 yrs.

SECONDARY OUTCOMES:
To investigate the risk of CVD and new onset diabetes in patients treated with specific types of ACEi or candesartan for hypertension | Time to first CV event calculated as the time (in days) between date of index prescription and date of the first registration of a CV event. Patients will be followed for min. 1 wk and up to 9 yrs (1999-2007). Median follow up time is estimated to 2 yrs.
To investigate the risk of hypertensive organ damage, renal failure and hyperlipidemia for patients treated with ACEi or candesartan | Time to first CV event calculated as the time (in days) between date of index prescription and date of the first registration of a CV event. Patients will be followed for min. 1 wk and up to 9 yrs (1999-2007). Median follow up time is estimated to 2 yrs.
Evaluate differences in use of health care resources, and assess the potential long term cost effectiveness | Differences in health care consumption will be estimated through models incorporating normalised costs, level of care, age, gender and study year

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Lindarck, Study Director — AstraZeneca Nordic
Locations (56):
- Sweden (56):
  - Research Site, Avesta
  - Research Site, Älvdalen
  - Research Site, Ängelholm
  - Research Site, Åkersberga
  - Research Site, Bengtsfors
  - Research Site, Borlänge
  - Research Site, Falun
  - Research Site, Farsta
  - Research Site, Fritsla
  - Research Site, Gagnef
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Grängesberg
  - Research Site, Grycksbo
  - Research Site, Hallstahammar
  - Research Site, Hägersten
  - Research Site, Hässelby
  - Research Site, Hedemora
  - Research Site, Helsingborg
  - Research Site, Henån
  - Research Site, Höllviken
  - Research Site, Jarfalla
  - Research Site, Kil
  - Research Site, Kolbäck
  - Research Site, Kolsva
  - Research Site, Köping
  - Research Site, Leksand
  - Research Site, Lidköping
  - Research Site, Likenäs
  - Research Site, Limhamn
  - Research Site, Ludvika
  - Research Site, Malmo
  - Research Site, Malung
  - Research Site, Mora
  - Research Site, Munka-Ljungby
  - Research Site, Norberg
  - Research Site, Sala
  - Research Site, Säter
  - Research Site, Skanör
  - Research Site, Skepplanda
  - Research Site, Skinnskatteberg
  - Research Site, Skogås
  - Research Site, Skoghall
  - Research Site, Skövde
  - Research Site, Skultuna
  - Research Site, Smedjebacken
  - Research Site, Stockholm
  - Research Site, Stora Höga
  - Research Site, Sunnansjö
  - Research Site, Sunne
  - Research Site, Svärdsjö
  - Research Site, Trollhättan
  - Research Site, Upplands Vasby
  - Research Site, Uppsala
  - Research Site, Vansbro
  - Research Site, Västerås

REFERENCES:
- [Derived] Hasvold LP, Bodegard J, Thuresson M, Stalhammar J, Hammar N, Sundstrom J, Russell D, Kjeldsen SE. Diabetes and CVD risk during angiotensin-converting enzyme inhibitor or angiotensin II receptor blocker treatment in hypertension: a study of 15,990 patients. J Hum Hypertens. 2014 Nov;28(11):663-9. doi: 10.1038/jhh.2014.43. Epub 2014 Jun 26. PMID 25211055